CLINICAL TRIAL: NCT06413420
Title: SUNOSI® (Solriamfetol) Pregnancy Registry: An Observational Study on the Safety of Solriamfetol Exposure in Pregnant Women and Their Offspring
Brief Title: SUNOSI® (Solriamfetol) Pregnancy Registry
Status: Recruiting | Type: Observational
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: JZP110-402
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Narcolepsy; Obstructive Sleep Apnea; Pregnant Women and Their Offspring
Keywords: Solriamfetol; SUNOSI; Axsome; Narcolepsy; Obstructive Sleep Apnea; Non-stimulant therapy; Dopamine norepinephrine reuptake inhibitor; Pregnancy outcomes; Infant outcomes
MeSH Terms: conditions — Narcolepsy; Sleep Apnea, Obstructive | interventions — solriamfetol; Central Nervous System Stimulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cohort 1: Solriamfetol-exposed participants with narcolepsy or OSA: Pregnant women with a diagnosis of narcolepsy or OSA
  Interventions: Drug: Sunosi (solriamfetol)
- Cohort 2: Unexposed participants with narcolepsy or OSA: Pregnant women with a diagnosis of narcolepsy or OSA
  Interventions: Other: No treatment
- Cohort 3: Other-exposed participants with narcolepsy or OSA: Pregnant women with a diagnosis of narcolepsy or OSA
  Interventions: Drug: Other prescription wake-promoting medications or stimulants
- Cohort 4: Solriamfetol-exposed participants without narcolepsy or OSA: Pregnant women without a diagnosis of narcolepsy or OSA
  Interventions: Drug: Sunosi (solriamfetol)
- Cohort 5: Other-exposed participants without narcolepsy or OSA: Pregnant women without a diagnosis of narcolepsy or OSA
  Interventions: Drug: Other prescription wake-promoting medications or stimulants

INTERVENTIONS:
Drug: Sunosi (solriamfetol) — Exposure to at least 1 dose of solriamfetol at any time during pregnancy.
  Groups: Cohort 1: Solriamfetol-exposed participants with narcolepsy or OSA; Cohort 4: Solriamfetol-exposed participants without narcolepsy or OSA
Drug: Other prescription wake-promoting medications or stimulants — Exposure to at least 1 dose of a prescription wake-promoting medication or stimulant at any time during pregnancy.
  Groups: Cohort 3: Other-exposed participants with narcolepsy or OSA; Cohort 5: Other-exposed participants without narcolepsy or OSA
Other: No treatment — No treatment
  Groups: Cohort 2: Unexposed participants with narcolepsy or OSA

SUMMARY:
The SUNOSI (solriamfetol) Pregnancy Registry is a prospective, multi-country, observational study to evaluate the safety of solriamfetol exposure during pregnancy in women with a diagnosis of narcolepsy or obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
The goal of the registry is to provide information on the safety of solriamfetol during pregnancy so that patients and physicians can weigh the benefits and risks of exposure during pregnancy and make informed treatment decisions.

The study collects health information from enrolled pregnant women and their healthcare providers related to their pregnancies and developing babies up to 1 year of age. The registry is strictly observational. Only data that are routinely documented in patients' medical records during the course of usual care will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women of any age
* Diagnosed with narcolepsy or obstructive sleep apnea OR has taken solriamfetol or other wake promoting medications or stimulants during pregnancy
* Resident of a country where solriamfetol is available for the treatment of excessive daytime sleepiness (EDS) associated with narcolepsy or OSA
* Provides written informed consent to participate in the study
* Authorization for her HCP(s) to provide data to the registry

Exclusion Criteria:

* Occurrence of pregnancy outcome prior to first contact with the registry coordination center (RCC)
* Inclusion of a prior pregnancy in the main analysis population

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include pregnant women of any age who reside in a country where solriamfetol is available for the treatment of narcolepsy or OSA, provide consent to participate as well as medical releases for their healthcare providers (HCPs) to provide data to the registry, and meet the criteria for inclusion into 1 of the 5 cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 1731 (Estimated)
Dates: Start 2019-07-31 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Long-term Safety | Baseline up to 12 months after pregnancy outcome

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Evidera, a PPD business unit, Morrisville, North Carolina
  - PPD, Inc., Wilmington, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com
- See also: Sunosi Pregnancy Registry Recruitment Website — https://sunosipregnancyregistry.com